CLINICAL TRIAL: NCT02593227
Title: A Randomized Multicenter Phase II Trial to Evaluate the Safety and Immunogenicity of Two Doses of Vaccination With Folate Receptor Alpha Peptides With GM-CSF in Patients With Triple Negative Breast Cancer Defined as Primary Tumor That is Her2-neu and Low (< 10%) ER/PR Nuclear Staining
Brief Title: Folate Receptor Alpha Peptide Vaccine With GM-CSF in Patients With Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marker Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRV-002
Record Dates: First submitted 2015-10-27; First posted 2015-11-02 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: TNBC
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose FRα vaccine (Experimental): FRα peptide vaccine with GM-CSF adjuvant - single ID administration - monthly vaccinations repeated 6 times followed by boosters every 6 months until recurrence
  Interventions: Biological: Low dose FRα vaccine
- High dose FRα vaccine (Experimental): FRα peptide vaccine with GM-CSF adjuvant - triple ID administration - monthly vaccinations repeated 6 times followed by boosters every 6 months until recurrence
  Interventions: Biological: High dose FRα vaccine
- Low dose FRα vaccine + cyclophosphamide (Experimental): Cyclophosphamide 300 mg/sqm as a 1 hour IV infusion 3 days prior to first vaccination. Followed by FRα peptide vaccine with GM-CSF adjuvant - ID administration - monthly vaccinations repeated 6 times followed by boosters every 6 months until recurrence
  Interventions: Biological: Low dose FRα vaccine; Drug: Cyclophosphamide
- High dose FRα vaccine + cyclophosphamide (Experimental): Cyclophosphamide 300 mg/sqm as a 1 hour IV infusion 3 days prior to first vaccination. Followed by FRα peptide vaccine with GM-CSF adjuvant - ID administration - monthly vaccinations repeated 6 times followed by boosters every 6 months until recurrence
  Interventions: Drug: Cyclophosphamide; Biological: High dose FRα vaccine

INTERVENTIONS:
Biological: Low dose FRα vaccine — 165ug per peptide ID injection
  Other Names: TPIV200
  Arms: Low dose FRα vaccine; Low dose FRα vaccine + cyclophosphamide
Drug: Cyclophosphamide — IV infusion over 1 hour
  Other Names: Cytoxan
  Arms: High dose FRα vaccine + cyclophosphamide; Low dose FRα vaccine + cyclophosphamide
Biological: High dose FRα vaccine — 500ug per peptide ID injection
  Other Names: TPIV200
  Arms: High dose FRα vaccine; High dose FRα vaccine + cyclophosphamide

SUMMARY:
This Phase II trial evaluates the safety and immunogenicity of two doses of the Folate Receptor Alpha (FRα) peptide vaccine mixed with GM-CSF as a vaccine adjuvant, with or without a immune priming with cyclophosphamide, as a consolidation therapy after neoadjuvant or adjuvant treatment of patients with Stage IIb-III triple negative breast cancer (TNBC).

DETAILED DESCRIPTION:
Triple negative breast cancers (TNBCs) occur in approximately 20-25% of all patients with breast cancer and are associated with a poor prognosis. Patients with TNBCs derive no benefit from targeted therapies. Excluding those patients who demonstrate a pathologic complete response following neoadjuvant chemotherapy, which is a minor fraction (i.e. 15%), overall survival is only 45% at 7 years.

Following standard of care, there are windows of opportunity to further and safely treat patients to prevent recurrence. Stimulating the immune system to produce T cells immunity specific for tumor antigens may significantly delay recurrence and cure patients.

The proposed vaccine is intended to induce T cells to survey for the reemergence of TNBCs and to prevent recurrence in the adjuvant setting. The vaccine strategy is antigen-specific and targets the Folate Receptor Alpha (FRα). FRα is an ideal target because of its limited expression in the healthy tissues and it high expression in 86% of TNBCs. Studies have shown that it is a biologically important marker that is associated with poorer clinical outcome and is retained in metastatic lesions.

The FRα vaccine include a pool of 5 peptides that are immunogenic epitopes and safely generate tissue-surveying CD4 T cell immune responses in patients tested in a recently completed phase I clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient, age 18 years or older;
2. Completely resected unilateral or bilateral primary carcinoma of the breast
3. Written informed consent must be obtained and documented according to the local regulatory requirements prior to beginning specific protocol procedures;
4. Primary tumor was negative for ER, PR (cut-off for positivity is >10% positive tumor cells with nuclear staining) and negative for Her2-neu (0 or 1+ on immunohistochemistry and/or normal gene copy number by in-situ hybridization); Central review is not required.
5. Completed primary treatment (surgery and radio/chemotherapy in adjuvant and/or neo-adjuvant setting) <360 days prior to first vaccination.
6. Completed last cycle of chemotherapy or radiation > 60 days prior to first vaccination
7. Either clinical or pathological Stage I (T1c), II, or III according to AJCC 7th edition

   * Note that patients with (i) non-invasive breast cancer (DCIS) alone, (ii) incidental (microscopic) nodal cancer without a primary tumor (pN1mi), or (iii) metastatic disease are excluded.
   * Resected tumor: No evidence of gross tumor at the surgical resection margin noted in the final surgery report. No evidence of gross residual adenopathy
8. Karnofsky index >= 70%;
9. Life expectancy of at least 5 years, disregarding the diagnosis of cancer;
10. Adequate Blood, renal and hepatic function, as determined within 28 days from registration:

    * ANC ≥ 1,500 / mm3
    * Platelet ≥ 100,000 / uL
    * Hgb > 9 g/dL
    * Creatinine ≤ 1.5 x ULN or 24-hour urine < Grade 2
    * Urinalysis with < 2+ proteinuria
    * Serum albumin ≥ 3 g/dL
    * SGOT (AST) ≤ 3 x ULN
11. Anti-nuclear antibody (ANA) negative or low-positive institutional range, as determined within 28 days from registration. Intermediate values (usually defined by a titer of ≤1:80, or as indicated by institutional range) are acceptable if there are, in the opinion of the Investigator, no early signs of an autoimmune disease.
12. Primary tumor is available for shipment to central laboratory for analysis of FRα expression by IHC.
13. Patients must be, in the opinion of the Investigator, available and compliant for treatment and follow-up.

Exclusion Criteria:

1. Clinical evidence of distant metastases per practice guidelines for breast cancer;
2. Inflammatory breast cancer or tumor with deep adherence or cutaneous invasion;
3. Known hypersensitivity reaction to the GM-CSF adjuvant; Any known contra-indication to GM-CSF or Cyclophosphamide treatment;
4. Pregnant or lactating patients. Patients of childbearing potential must have a negative pregnancy test (urine or serum) within 7 days prior to registration and must implement adequate contraceptive measures during study treatment;
5. Active autoimmune disease requiring therapy within the past 2 years (Note: patients with vitiligo, Grave's disease or psoriasis not requiring systemic treatment within the past 2 years are not excluded);
6. Other uncontrolled illness or medical condition, such as active infection, symptomatic heart failure (New York Heart Association class III or IV; moderate to severe objective evidence of cardiovascular disease), unstable angina pectoris, myocardial infarction or stroke within last 6 months, psychiatric illness that may limit compliance with study requirement or interfere with the understanding and giving of informed consent;
7. Prior active secondary malignancy < 5 years prior to consent (except non-melanomatous skin cancer or carcinoma in situ of the uterine cervix) or currently receiving other specific treatment for this cancer (including monoclonal antibody or pathway inhibitor);
8. Completed treatment with systemic corticosteroid or immune-modulators < 30 days prior to registration;
9. Planned treatment with other experimental drugs or any other non-hormonal anti-cancer therapy;
10. Immunocompromised patients, including patients with known HIV infection;
11. Symptomatic thyroid disease, unless negative for thyroid antibodies (TSH receptor, TPO, thyroglobulin).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Immune response | 3 years
  Emergence of B and T cell immunity targeting the folate receptor alpha

SECONDARY OUTCOMES:
Folate receptor alpha expression | Baseline
  To determine FRα expression status of primary tumors
Relapse Free Survival | 3 years
  RFS in relation to FR specific immune response
Safety and tolerability (treatment emergent adverse events and injection site reactions) | 3 years
  Incidence of treatment emergent adverse events and injection site reactions

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kenney, MD, Study Director — Marker Therapeutics, Inc.
Locations (11):
- United States (11):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Maryland - Greenebaum Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Center, Detroit, Michigan
  - MidAmerica Division,Inc, Kansas City, Missouri
  - The Valley Hospital, Paramus, New Jersey
  - Mount Sinai Hospital, New York, New York
  - Montefiore Medical Center, Einstein Cancer Center, New York, New York
  - Oncology Hematology Care, Cincinnati, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology Presbyterian Cancer Center Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Corporate website — http://www.markertherapeutics.com